CLINICAL TRIAL: NCT00138411
Title: Randomized, Placebo-Controlled, Double Blind, Dose-Escalation Phase I Study of the Safety, Tolerability, and Pharmacokinetics of a Single Intravenous Dose of ETI-204 [Anthim(TM)] and Its Potential Interaction With Ciprofloxacin
Brief Title: Monoclonal Antibody for Treatment of Inhalation Anthrax
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 04-096; AH-101
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2006-07

CONDITIONS: Bacillus Anthracis (Anthrax)
Keywords: anthrax, Bacillus anthracis, monoclonal antibody, ETI-204
MeSH Terms: conditions — Anthrax | interventions — Ciprofloxacin; obiltoxaximab

INTERVENTIONS:
Drug: Ciprofloxacin 500 mg
Drug: ETI-204 (Anthim)

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics (how long a drug stays in the bloodstream and how high the levels of the drug are at different times) of ETI-204 following intravenous (IV-into a vein) injections, and to evaluate the effects that ETI-204 may have on the pharmacokinetics of oral (by mouth) ciprofloxacin, an antibiotic approved by the U.S. Food and Drug Administration (FDA). ETI-204 is an experimental drug (not approved by the FDA) intended to protect against anthrax (a bacterial infection). Approximately 36 male and female healthy volunteers ages 18 to 50 will be in this study. Participation in this study may last up to eight weeks. Volunteers will have a single IV dose of the ETI-204 study drug or placebo (inactive substance, and some participants will also receive ciprofloxacin. They will stay in the Clinical Pharmacology Unit at least 36 hours after the dose.

DETAILED DESCRIPTION:
This initial study with ETI-204 will examine the safety and pharmacokinetics of ETI-204 following IV administration both in the absence and presence of ciprofloxacin. The pharmacokinetics of ciprofloxacin in the presence of ETI-204 will also be determined. This study is a placebo-controlled, double-blind, randomized study which will be conducted at a single site. Healthy male and female volunteers will be recruited from the Columbus, OH area, and will have a maximum participation period of 7 months for each subject (from enrollment to end of follow-up period). The study population will roughly parallel the ethnicity of this geographic area. Because this is the first time that ETI-204 is studied in man, individuals under the age of 18 will not be permitted to participate in the study. Part 1 is a randomized, placebo-controlled, double-blind study being conducted at a single study site. Part 2 will be double-blind with respect to ETI-204 but not blinded for oral ciprofloxacin. Part 1 of the study is the dose escalation portion, in which the safety, tolerability, and pharmacokinetics of single IV doses of ETI-204 will be evaluated. Three dose levels are proposed for study: 18 mg, 54 mg, and 108 mg. At each dose level, 3 males and 3 females will be randomly assigned to active drug and 1 male and 1 female will be randomly assigned to placebo. Thus, at least 24 subjects will be studied in Part 1. Part 2 of the study will determine the safety, tolerability and pharmacokinetics of a single IV dose (108 mg dose from part 1, presuming no safety or tolerability issues), and whether or not there is an effect of ETI-204 on ciprofloxacin pharmacokinetics. There will be 2 groups of 6 subjects each. The first cohort will receive ETI-204 plus ciprofloxacin and the second will receive ETI-204 placebo plus ciprofloxacin. Together with the comparable group from part 1, this will allow the determination of the effects of ciprofloxacin on ETI-204 pharmacokinetics and of ETI-204 on ciprofloxacin pharmacokinetics. Subjects will receive ciprofloxacin 500 mg or placebo every 12 hours for a total of 14 days beginning at the time of ETI-204/placebo administration. It is anticipated that the number of subjects in part 1 of the study (18 receiving active ETI-204 and 6 receiving placebo) will be sufficient to allow a preliminary assessment of safety and efficacy (ETI-204 concentration). In part 2, 12 subjects will receive active ETI-204 (108 mg dose from part 1, presuming no safety or tolerability issues). Of these, 6 will also receive oral ciprofloxacin and 6 will serve as the controls (i.e., ETI-204 alone). An additional cohort of 6 subjects will receive ETI-204 placebo and oral ciprofloxacin. This number of subjects should be sufficient to provide an indication of the presence of a drug-drug interaction between ETI-204 and ciprofloxacin, but not necessarily the magnitude. All statistical comparisons will be performed using two sided tests at an alpha level of 0.05 unless specifically stated otherwise. All statistical null hypotheses assert that there are no differences between treatments. Because this is the first study in man with ETI-204, the full risks can not be determined. ETI-204 is being tested for its utility in preventing the life-threatening sequelae that may occur following exposure to anthrax. The results of this study could demonstrate that ETI-204 has an acceptable safety profile and that it has a pharmacokinetic profile that will provide for serum concentrations of the drug (antibody) over time that will be effective in preventing the toxicity of one of the exotoxins produced by B. anthracis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects between the ages of 18-50 inclusive at the time of enrollment. In each of the drug cohorts (subgroups), at least two of the subjects must be female.
2. The following screening laboratory parameters must be within the normal range: AST, ALT, alkaline phosphatase, hemoglobin, and serum creatinine. No repeat testing is allowed for these analytes. For any other clinical chemistry analyte or CBC (including differential and platelet count) parameter that is outside the normal range, the PI and the sponsor's medical monitor will confer and must agree in writing that the value has no clinical significance before the subject will be allowed to enter the study.
3. The values for the following tests at screening are to be:

   G-6-P dehydrogenase - normal HBsAG - negative HBV - negative Anti-HCV - negative Anti-HIV (HIV antibody test) - negative Urine drug screen (including cotinine) - negative
4. Female subjects of childbearing potential must agree to practice abstinence or to use a licensed, effective form of birth control (e.g., oral contraceptives, diaphragm or condom in combination with contraceptive jelly, cream or foam, intrauterine contraceptive device, Depo-Provera®, skin patch, vaginal ring, or cervical cap) for at least 30 days prior to enrollment and for the duration of the study, including the follow-up period. Females using hormonal contraceptives must agree to use at least one other method for at least 30 days prior to enrollment and for the duration of the study, including the follow-up period.
5. Female subjects must have a negative pregnancy test.
6. No history of hospitalization for illness within the six months prior to study enrollment.
7. Non-smoker or ex-smoker. If a subject is an ex-smoker, he/she must not have used nicotine for at least 6 months prior to enrollment. This will be confirmed by a negative urine test for cotinine.
8. Able to spend the two days specified in the study schedule confined in a facility under study rules.
9. Able to read, understand and sign the Informed Consent form.

Exclusion Criteria:

1. Routine consumption of any medication (prescription or OTC), vitamin, mineral, antacid, or dietary supplement, for one week before and during the study. The sole exception are hormonal contraceptive agents, as detailed above, hormone replacement therapy, and thyroid replacement therapy. Subjects must be specifically reminded that antacids are excluded.
2. Blood pressure greater than 145 mm Hg systolic and 95 mm Hg diastolic.
3. Contraindication to the use of ciprofloxacin or any quinolone. (Part 2 only).
4. Contraindication to the use of any monoclonal antibody.
5. Medical condition that in the Investigator's opinion could adversely impact the subject's participation, safety or conduct of the study.
6. Subject has taken an investigational medication in the previous three months.
7. The subject has a history of drug or alcohol abuse within the past two years.
8. The subject is female and plans to become pregnant during the study or the 42 day follow-up period.
9. Calculated Body Mass Index (BMI) greater than 35 or less than 18.5.
10. The subject has been previously vaccinated with anthrax or has participated in clinical research involving anthrax.
11. Any EKG abnormality except for the following:

    1. Sinus bradycardia in younger, athletic subjects
    2. Mild first degree A-V block (P-R interval < 0.23 sec)
    3. Mild right or left axis deviation
    4. Incomplete right bundle branch block DMID does not allow for exceptions of eligibility criteria waivers for enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36
Dates: Start 2005-10; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States